CLINICAL TRIAL: NCT02612220
Title: Effectiveness of BioFoam® Surgical Matrix to Improve Hemostasis During Liver Resection - A Randomized Controlled Trial
Brief Title: Effectiveness of BioFoam® Surgical Matrix to Improve Hemostasis During Liver Resection
Acronym: BioFoam
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Technische Universität Dresden (Other)
Collaborators: CryoLife, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: VTG-03
Record Dates: First submitted 2015-11-13; First posted 2015-11-23 (Estimated); Last update posted 2017-10-20 (Actual); Status verified 2017-01

CONDITIONS: Hemorrhage
Keywords: liver resection
MeSH Terms: conditions — Hemorrhage

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Experimental Group (Experimental): Complete hemostasis will be achieved using BioFoam® Surgical Matrix
  Interventions: Procedure: BioFoam® Surgical Matrix
- Control Group (Active Comparator): Complete hemostasis will be achieved without the use of topical agents, using conservative hemostasis
  Interventions: Other: Conservative hemostasis

INTERVENTIONS:
Procedure: BioFoam® Surgical Matrix — Complete hemostasis is achieved by direct application of BioFoam® (Cryolife Inc., Kennesaw, GA) to the transection surface area of the liver. In addition, the surgeon may use conventional methods such as argon beam coagulation and warm sponges. If more than one syringe of BioFoam® is required to cover the entire transection surface area, a second syringe maybe used. BioFoam® Surgical Matrix will be used according to the supplier's instructions.
  Arms: Experimental Group
Other: Conservative hemostasis — Complete hemostasis will be achieved without the use of topical agents
  Arms: Control Group

SUMMARY:
The present randomized controlled trial evaluates the efficacy and safety of BioFoam® Surgical Matrix in patients undergoing elective liver resection. In contrast to other topical agents, the surgical adhesive BioFoam® Surgical Matrix may not only accelerate hemostasis but also facilitate sealing of bile ducts and thus has the potential to reduce the incidence of postoperative complications.

The primary objective of this trial is to show that time-to-complete hemostasis can be reduced using BioFoam® Surgical Matrix as compared to the conventional approach.

DETAILED DESCRIPTION:
Hepatic resection is the primary therapy for various hepatobiliary disorders. Advances in preoperative imaging, surgical technique, and perioperative management have markedly improved outcomes and extended the indications for hepatic resection within the past three decades. However, liver resection remains associated with substantial morbidity and mortality of up to 60% and 10%, respectively. The outcome of patients undergoing hepatic resection is closely linked to the amount of intraoperative blood loss. Hemorrhage from the resection surface contributes significantly to the amount of blood loss. In addition, bile leakage from the resection surface presents a persistent clinical challenge. In fact, bile leakage remains the most frequent complication after hepatic resection with an incidence of 5 - 25%. Various topical agents have so far been suggested to facilitate hemostasis with the ultimate aim to improve perioperative outcome. However, none of these agents has so far gained wide acceptance, possibly due to their impractical method of application. Furthermore, these 'hemostatic agents' have been primarily designed to improve hemostasis and showed no effect on perioperative complications and in particular the incidence of bile leakage.

The present randomized controlled trial evaluates the efficacy and safety of BioFoam® Surgical Matrix in patients undergoing elective liver resection. In contrast to other topical agents, the surgical adhesive BioFoam® Surgical Matrix may not only accelerate hemostasis but also facilitate sealing of bile ducts and thus has the potential to reduce the incidence of postoperative complications.

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled for elective hepatic resection
* Age equal or greater than 18 years
* Informed consent

Exclusion Criteria:

* Previous treatment with BioFoam® Surgical Matrix
* Known sensitivity to materials of bovine origin
* Known sensitivity to glutaraldehyde
* Abnormal calcium metabolism (e.g. chronic renal failure, hyperparathyreoidism)
* Minimally invasive procedure planned
* Impaired mental state or language problems
* Expected lack of compliance

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 101 (Actual)
Dates: Start 2015-12-03 (Actual); Primary Completion 2017-09-06 (Actual); Study Completion 2017-09-06 (Actual)

PRIMARY OUTCOMES:
Time-to-complete hemostasis | 3 minutes

CONTACTS AND LOCATIONS:
Overall Officials: Christoph Reißfelder, MD, Principal Investigator — Department of Visceral, Thoracic and Vascular Surgery, University Hospital Carl Gustav Carus, TU Dresden, Germany
Locations (1):
- Department of Visceral, Thoracic and Vascular Surgery, University Hospital Carl Gustav Carus, TU Dresden, Germany, Dresden, Saxony, Germany

REFERENCES:
- [Derived] Rahbari NN, Birgin E, Sturm D, Schwanebeck U, Weitz J, Reissfelder C. Randomized clinical trial of BioFoam(R) Surgical Matrix to achieve hemostasis after liver resection. HPB (Oxford). 2020 Jul;22(7):987-995. doi: 10.1016/j.hpb.2019.10.1529. Epub 2019 Nov 1. PMID 31680010